CLINICAL TRIAL: NCT03781102
Title: Type 2 Diabetes Prevention in Community Health Care Settings for at Risk Children and Mothers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Melanie Hingle, Assistant Professor, Department of Nutritional Sciences, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R34DK118486-01 (NIH)
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: PreDiabetes; Type 2 Diabetes
Keywords: Type 2 Diabetes; Diabetes Prevention; Prediabetes Intervention; Mothers; Children; Federally Qualified Health Center (FQHC) Program
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants (60 children and their biological mothers (n=120)) will be assigned to a clinic location nearest to their home address, which will determine the order in which they will complete the 16-week intervention. Two clinics were selected to participate in this pilot study. Randomization to the intervention and wait-list control conditions will be performed *by site* (flip of a coin). Randomization by site is proposed as it has the least potential for contamination during the initial delivery period. Group A participants (n=30) will begin the 16-week face-to-face group program immediately, whereas the Group B participants (n=30) will receive normal standard of care. After 16 weeks, the Group A participants will transition to follow-up while the Group B participants begin the intervention. This design is responsive to standards of care for T2D prevention by primary care providers and will provide the opportunity to investigate all the outcome questions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Arm 1, or intervention participants (n=60), will participate in a 16-week face-to-face diabetes prevention group program '16-Week Diabetes Prevention Program for Mothers and Children' and then will transition to a 16-week follow-up period.
  Interventions: Behavioral: 16-Week Diabetes Prevention Program for Mothers and Children
- Wait-listed Control (Other): Arm 2, or wait-listed controls (n=60), will receive the typical standard of care during the first 16-weeks, followed by the 16-week face-to-face group diabetes prevention program '16-Week Diabetes Prevention Program for Mothers and Children'.
  Interventions: Behavioral: 16-Week Diabetes Prevention Program for Mothers and Children

INTERVENTIONS:
Behavioral: 16-Week Diabetes Prevention Program for Mothers and Children — The 16-week intervention is focused on ways to modify behaviors associated with the pathogenesis of Type 2 Diabetes in youth, while engaging participants in fun, active, and interactive food demonstrations, energy balance, and physical activities appropriate for all the family. Weekly sessions will consist of: (1) physical activity upon arrival; (2) small group discussions; (3) hands-on food preparation and tasting opportunities; (4) low- to no-cost fun family physical activities; (5) energy balance activities (e.g. label reading) to increase foundational knowledge; and, (6) opportunities to set new weekly goals.

SUMMARY:
The two main questions that this research study will answer:

1. will a 16-week community-based diabetes prevention program for delivery to at-risk mothers and children in a Federally Qualified Health Center (FQHC) setting show (a) pre- and post-intervention improvements to Type 2 Diabetes risk factors in 60 mother-child dyads; (b) intervention vs. control improvements to T2D risk factors in 30 mother-child dyads; and (c) maintenance effects to changes to Type 2 Diabetes risk factors in 30 mother-child dyads; and
2. based on the acceptability, adoption, relevance to FQHC and participants, feasibility, fidelity, program costs, and factors influencing sustainability of this program, can it be disseminated nationwide to other FQHC's?

The investigators hypothesize that participants (a) will show improvements following the intervention to T2D risk factors, (b) in the intervention will show significant improvements to T2D risk factors in versus the controls, and (c) will maintain the benefits beyond the 16-week intervention. The investigators also predict that this program will meet criteria to be disseminated nationwide to other FQHC's.

DETAILED DESCRIPTION:
The goal is to implement and evaluate the effects of a 16-week behavioral lifestyle intervention on Type 2 Diabetes (T2D) risk factors delivered by trained staff at a Federally Qualified Health Center (FQHC) to 60 mothers with prediabetes or a history of gestational diabetes (GDM) and 60 overweight/obese children. The specific aims are to (1) adapt an efficacious community-based diabetes prevention program for delivery to FQHC patients, (2) evaluate indicators of program implementation and potential for dissemination (Proctor 2011), and (3) assess the preliminary impact of the program on participants' T2D risk factors.

The study aims to adapt an efficacious community-based diabetes prevention program developed for delivery to at-risk mothers and children at a FQHC. Successful T2D prevention in children necessitates family adoption of lifestyle behaviors associated with prevention of excess weight gain, while supporting normal growth and development. In accord with the 2012 Institute of Medicine Report (IOM 2012) and guidelines set forth by an Expert Committee (Barlow 2007), three healthy lifestyle goals form the basis for youth-focused aspects of the intervention: i) make physical activity an integral and routine part of life; ii) eat a healthy diet (both quality and quantity), and, iii) create food and physical activity environments to insure healthy options and behaviors are the routine, easy choice. These goals align with two evidence-based T2D prevention goals mothers will be encouraged to adopt: i) lose 7% of body weight through healthy eating, and ii) participate in at least 150 minutes of moderate-to-vigorous physical activity each week. Achievement of these goals has been associated with significant T2D risk reduction in participants of programs based on the Centers for Disease Control and Prevention (CDC) National Diabetes Prevention Program (CDC 2017, Albright 2013). The intervention duration, content, and activities, designed to support families in meeting these recommendations, were drawn from the intervention literature (Wilfley 2010, Epstein 2007, Ackermann 2008, Hingle 2015). Intervention "dose" (duration × time) was modeled after the successful adult-focused DPP/YDPP (characterized by 16 core sessions) and the recently released 2017 U.S. Preventive Services Task Force (USPSTF) evidence-based recommendations for weight loss, behavior change, and cardio-metabolic risk reduction in youth (O'Connor 2017). The topics are focused on practical, culturally-relevant strategies for modifying the behaviors associated with the pathogenesis of T2D in youth (Spruijt-Metz 2014) (e.g., availability and accessibility of nutrient- and calorie-dense foods and food preparation strategies in the home, reducing intake of sugar-sweetened beverages, increasing time spent in physical activity/decreasing time spent in sedentary activities, stress management, and obtaining quality sleep), while engaging participants in fun, active, and interactive food demonstrations, energy balance, and physical activities appropriate for the entire family. All sessions are group-based (attended by up to 10 families total) and led by a minimum of two trained bilingual FQHC health and wellness staff. The sessions will be approximately 1.5-2 hours in length and conducted over 16 consecutive weeks at one of two FQHC locations. The sessions foster skill building and provide repeated opportunities to practice healthy lifestyle behaviors. Each session will follow a similar format consisting of: (1) a featured physical activity encouraging families to get moving upon arrival; (2) small group discussions focused on goal-setting and building intra- and inter-family camaraderie; (3) hands-on food preparation and tasting opportunities centered around vegetables, whole grains, and legumes; (4) low- to no-cost fun family physical activities (on alternating weeks, mothers will participate in a moderated discussion on proactive parenting); (5) energy balance activities (e.g. label reading) to increase foundational knowledge and skills related to healthy food selection, physical activity benefits, and creating a supportive home environment; and, (6) opportunities to set new weekly goals (or revise previous goals).

The second aim evaluates program implementation outcomes including acceptability, adoption, relevance to FQHC and participants, feasibility, fidelity, program costs, and factors influencing sustainability. Consistent with the tenets of implementation science (Glasgow 2012), these variables are assessed at recommended time points (Proctor 2011) to insure all aspects of the intervention work as intended, including participant acceptability (participant satisfaction) and relevance to FQHC personnel and study participants (rated using brief surveys of the relevance of the intervention to daily life, promoters and barriers to program attendance and engagement, the degree to which families report using the intervention to guide behavioral choices, and surveys of lifestyle coaches trained to deliver the intervention). The investigators also assess adoption by the FQHC and integration with the existing clinical setting (ascertained through semi-structured interviews with FQHC wellness staff and administrators exploring 'fit' among existing program offerings, availability of personnel and resources needed to implement, and potential for reimbursement) and feasibility (of delivery by providers and FQHC determined by recruitment, enrollment, and retention rates, adherence data including session attendance and observed participant engagement with intervention activities; a brief, three-question interview will be conducted with every eligible respondent who elects not to participate). Fidelity is assessed through observation of research staff following an established rubric, and program costs are evaluated using a bottom-up micro-costing approach (for participants, surveys assessing cost, burden, and benefit such as time and resources spent in travel, services, equipment, and food to meet program recommendations; FQHC direct medical and non-medical costs including personnel gross hourly salaries, intervention material costs, and overhead costs related to use of facilities for prevention services are tracked and analyzed in partnership with FQHC data team members). The investigators also explore the potential for replication and dissemination using semi-structured interviews with the FQHC wellness staff assigned to coordinate and deliver the program, and administrators and advisory board members who understand how to align the intervention with the FQHC's fiscal and strategic plans, and who have relationships with other FQHCs in Arizona and nationally. Program sustainability is also of great interest to the FQHC, thus our a priori focus on factors influencing sustainability (e.g., reach, integration with other health/wellness programs, institutionalization) beyond the research funding period are a major consideration throughout the proposed study. At the conclusion of the proposed work, this evaluation is designed to produce an intervention curriculum and approach suitable for replication and scaling across a larger number of (cluster-randomized) FQHC sites.

The third aim is to assess the preliminary efficacy of the program on T2D risk factors including weight status, metabolic syndrome phenotype, lifestyle behaviors, and socio-environmental determinants of health outcomes in 60 mothers and 60 children participating in the 16-week intervention. Intervention participants are measured at Week 0 (baseline), Week 16 (post-intervention), and Week 32 (maintenance) and wait-listed control participants at Week 0 (baseline), Week 16 (follow-up and pre-intervention), and Week 32 (post-intervention). Measurements are conducted by trained research staff following standardized measurement procedures, and take place at the FQHC site to which the child and parent is assigned. Care is taken to avoid simultaneous scheduling of intervention and wait-listed control families.

ELIGIBILITY:
Inclusion Criteria:

Child:

8-12-years-old (if the mother has more than one child in the age range, the oldest child will be invited to participate; other children will be invited to join if the mother wishes it, but will not be measured),

overweight/obese (≥85th percentile of BMI for age and sex, and ≥2 of the following T2D risk factors: family history of T2D in first or second degree relative; or, identify as a racial/ethnic minority; or, exhibit signs of insulin resistance or conditions associated with insulin resistance, or mother with T2D or GDM during gestation.

Able to read and speak English, and provide written assent.

Mother:

18-54 years-old,

BMI ≥ 25 kg/m2 and a risk score ≥5 on the seven-item American Diabetes Association's Diabetes Risk Assessment (84). In addition, women must have prediabetes, determined by an HbA1c value >5.7% and <6.5%, or, a self-reported or chart documented history of gestational diabetes mellitus with an HbA1c <6.5% and/or casual capillary blood glucose <199 mg/dL.

Must be willing to participate with their child in all intervention activities and sessions,

Able to read and speak English or Spanish, and provide informed consent.

Exclusion Criteria:

Mother:

No evidence of prediabetes

Currently pregnant or planning to become pregnant during the study

Have any condition or use any medication that could alter glucose metabolism or weight

Have suffered a heart attack, stroke or transient ischemic attack (TIA) in the past 6 months

Have uncontrolled hypertension (systolic >180 mmHg or diastolic >105 mmHg)

Received treatment for cancer (excluding surgery alone) within the last 2 years (excluding skin cancer)

Report chest pain, shortness of breath with minimal activity or at rest or unexplained dizziness or fainting with physical activity,

Have chronic lung disease, chronic obstructive pulmonary disease, or asthma requiring home oxygen therapy,

Current use of anti-diabetes medications for the treatment of diagnosed diabetes, are unable to communicate with research staff (including intervention staff),

Do not have a child within the designated age range (8-12-years-old),

Unable to speak or read English or Spanish.

Ages: 8 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | Baseline, Week 16, Week 32
  Body weight (kg) is measured using a calibrated, Cardinal Detecto ProDoc Series PD300MHR Digital Physician scale and a Cardinal Detecto 758C Weight Indicator
Change in Body Height | Baseline, Week 16, Week 32
  Body height (cm) measured using a calibrated, Cardinal Detecto ProDoc Series PD300MHR Digital Physician scale with a mechanical height rod and a Cardinal Detecto 758C Weight Indicator with a Seca 213 Portable Stadiometer.
Change in Body Mass Index (BMI) | Baseline, Week 16, Week 32
  BMI (kg/m2) is categorized using international classifications of BMI (overweight, 25-29.9kg/m2; obese, >30kg/m2) (WHO 2006).
Change in Body Mass Index (BMI) Percentile | Baseline, Week 16, Week 32
  BMI percentile in children is determined using age- and sex-specific growth charts developed by the CDC in 2000 (Kuczmarski 2000).

SECONDARY OUTCOMES:
Change in Waist Circumference | Baseline, Week 16, Week 32
  Child and adult waist circumferences are measured at the umbilicus. All measures are completed in duplicate, and the average of the two measures is used.
Change in Blood Pressure | Baseline, Week 16, Week 32
  Blood pressure assessed with an aneroid sphygmomanometer and with a Mindray Accutorr V vital signs monitor with an appropriate-sized cuff after participants are seated and relaxed for at least 5 minutes.
Change in HbA1C | Baseline, Week 16, Week 32
  HbA1C as assessed using a finger stick sample will be collected using a Siemens Diagnostics DCA HbA1C analyzer.
Change in Total Cholesterol / HDL-cholesterol | Baseline, Week 16, Week 32
  Total Cholesterol and HDL-cholesterol as assessed using a finger stick sample will be measured using a Cholestech LDX® lipid analyzer.
Change in Dietary Intake (daily eating patterns) | Baseline, Week 16, Week 32
  Dietary Intake - Child - assessed with interviewer-administered 24-hr dietary recalls. Parent- assessed using Arizona Food Frequency Questionnaire (AFFQ).
Change in Moderate to vigorous physical activity (MVPA) and sedentary behavior | Baseline, Week 16, Week 32
  MVPA and sedentary behavior - Child - assessed using the Youth Activity Profile (YAP). Parent - assessed using the Arizona Activity Frequency Questionnaire (AAFQ).
Change in sleep behavior (daily sleeping patterns) | Baseline, Week 16, Week 32
  Sleep Behavior - Child - assessed using the Children's Sleep Habits Questionnaire, Abbreviated. Adult - N/A
Change in home food and physical activity environment | Baseline, Week 16, Week 32
  Home food and physical activity environment - assessed using the Family Nutrition and Physical Activity Tool (FNPA).
Change in demographic and social and environmental risk factors for T2D | Baseline, Week 16, Week 32
  Demographic and social and environmental risk factors for T2D will be assessed using the Sangre Por Salud Biobank Health Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie D Hingle, PhD, Principal Investigator — University of Arizona; David G Marrero, PhD, Principal Investigator — University of Arizona
Locations (1):
- El Rio Community Health Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Committee on Accelerating Progress in Obesity Prevention; Food and Nutrition Board; Institute of Medicine; Glickman D, Parker L, Sim LJ, Del Valle Cook H, Miller EA, editors. Accelerating Progress in Obesity Prevention: Solving the Weight of the Nation. Washington (DC): National Academies Press (US); 2012 May 8. Available from http://www.ncbi.nlm.nih.gov/books/NBK201141/ PMID 24830053
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Centers for Disease Control and Prevention. National Diabetes Prevention Program 2017. Available at: https://www.cdc.gov/diabetes/prevention/index.html [Accessed on October 18, 2017]
- [Background] Albright AL, Gregg EW. Preventing type 2 diabetes in communities across the U.S.: the National Diabetes Prevention Program. Am J Prev Med. 2013 Apr;44(4 Suppl 4):S346-51. doi: 10.1016/j.amepre.2012.12.009. PMID 23498297
- [Background] Wilfley DE, Vannucci A, White EK. Early intervention of eating- and weight-related problems. J Clin Psychol Med Settings. 2010 Dec;17(4):285-300. doi: 10.1007/s10880-010-9209-0. PMID 20960039
- [Background] Epstein LH, Paluch RA, Roemmich JN, Beecher MD. Family-based obesity treatment, then and now: twenty-five years of pediatric obesity treatment. Health Psychol. 2007 Jul;26(4):381-91. doi: 10.1037/0278-6133.26.4.381. PMID 17605557
- [Background] Ackermann RT, Finch EA, Brizendine E, Zhou H, Marrero DG. Translating the Diabetes Prevention Program into the community. The DEPLOY Pilot Study. Am J Prev Med. 2008 Oct;35(4):357-63. doi: 10.1016/j.amepre.2008.06.035. PMID 18779029
- [Background] Hingle MD, Turner T, Kutob R, Merchant N, Roe DJ, Stump C, Going SB. The EPIC Kids Study: a randomized family-focused YMCA-based intervention to prevent type 2 diabetes in at-risk youth. BMC Public Health. 2015 Dec 18;15:1253. doi: 10.1186/s12889-015-2595-3. PMID 26679186
- [Background] O'Connor EA, Evans CV, Burda BU, Walsh ES, Eder M, Lozano P. Screening for Obesity and Intervention for Weight Management in Children and Adolescents: Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2017 Jun 20;317(23):2427-2444. doi: 10.1001/jama.2017.0332. PMID 28632873
- [Background] Spruijt-Metz D, O'Reilly GA, Cook L, Page KA, Quinn C. Behavioral contributions to the pathogenesis of type 2 diabetes. Curr Diab Rep. 2014 Apr;14(4):475. doi: 10.1007/s11892-014-0475-3. PMID 24604714
- [Background] Glasgow RE, Vinson C, Chambers D, Khoury MJ, Kaplan RM, Hunter C. National Institutes of Health approaches to dissemination and implementation science: current and future directions. Am J Public Health. 2012 Jul;102(7):1274-81. doi: 10.2105/AJPH.2012.300755. Epub 2012 May 17. PMID 22594758
- [Background] World Health Organization (WHO). BMI classification. 2006 Available at: http://apps.who.int/bmi/index.jsp?introPage=intro_3.html [Accessed on October 18, 2017]
- [Background] Kuczmarski RJ, Ogden CL, Grummer-Strawn LM, Flegal KM, Guo SS, Wei R, Mei Z, Curtin LR, Roche AF, Johnson CL. CDC growth charts: United States. Adv Data. 2000 Jun 8;(314):1-27. PMID 11183293
- [Derived] Marrero DG, Blew RM, Palmer KNB, James K, Roe DJ, Hingle MD. Rationale and design of a type 2 diabetes prevention intervention for at-risk mothers and children at a Federally Qualified Healthcare Center: EPIC El Rio Families Study Protocol. BMC Public Health. 2021 Feb 12;21(1):346. doi: 10.1186/s12889-021-10392-w. PMID 33579240